CLINICAL TRIAL: NCT04654026
Title: Single-center, Prospective, Controlled Study of the Safety and Efficacy of Aspirin and Clopidogrel in Ischemic Cardiovascular and Cerebrovascular Patients Complications With CAA
Brief Title: the Safety and Efficacy of Antiplatelet Therapy in Patients of CAA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20200601034-FS01
Record Dates: First submitted 2020-10-11; First posted 2020-12-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-11

CONDITIONS: Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy | interventions — Aspirin; Clopidogrel; Ticagrelor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAA Group: Patients with cardiovascular and cerebrovascular disease with cerebral amyloidosis
  Interventions: Drug: Aspirin/Clopidogrel
- None CAA Group: Patients with cardio-cerebrovascular disease without cerebral amyloid vascular disease
  Interventions: Drug: Aspirin/Clopidogrel

INTERVENTIONS:
Drug: Aspirin/Clopidogrel — No intervention, only observational studies
  Other Names: ticagrelor

SUMMARY:
Ischemic cardiovascular and cerebrovascular diseases are the main causes of death among people. Antiplatelet threrapy is very important for patients to prevent ischemic cardiovascular and cerebrovascular diseases.Ischemic cardiovascular patients of cerebral amyloid angiopathy (CAA) patients is as high as 20%, aspirin and clopidogrel is applied to prevent or treat the patient with CAA is controversial, there is no valid evidence of CAA crowd is safe to use of antiplatelet drugs, but progress in clinical treatment is usually based on patient condition for antiplatelet agents to prevent the occurrence of adverse events, such as blood clots.Therefore, this study is intended to be a single-center, prospective study of patients with ischemic cardiovascular and cerebrovascular diseases taking aspirin and clopidogrel, to determine whether the patients are combined with CAA , and to conduct a follow-up study for 12 months after team inclusion:1) The prevalence rate and gene spectrum of ischemic cardiovascular and cerebrovascular diseases among CAA patients enrolled in our hospital were analyzed;2) To explore the correlation between aspirin and clopidogrel drug genes and blood drug concentrations and diseases in patients with ischemic cardiovascular and cerebrovascular diseases complicated with CAA;3) To evaluate the efficacy and safety of aspirin and clopidogrel in patients with ischemic cardiovascular and cerebrovascular diseases who combined with CAA.

DETAILED DESCRIPTION:
This project intends to observation of bleeding the application of antiplatelet in patients with CAA, so as to provide effective clinical evidence for the further application of clopidogrel and aspirin in patients with CAA in the future, and to provide reference basis for the accurate formulation of clinical treatment plans and the balance of health risks brought by adverse bleeding reactions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CAA
* Must be able to swallow tablets

Exclusion Criteria:

* Clopidogrel gene was non-CYP2C19 *1 patients.
* Patients with surgical thrombolysis .
* Patients with arteritis, aneurysms, arterial trauma and other risk factors were excluded.
* Patients with tumours, infections, fever, inflammatory diseases, post-embolization bleeding, peripheral vascular thrombosis or embolization, and other blood diseases such as hemophilia were excluded.
* Currently receiving treatment in another experimental device or drug study, or completing treatment in another experimental device or drug study ≤30 days.
* Patients are allergic to any of the ingredients known to be given aspirin or clopidogrel.
* Patients has an unstable medical condition, or is otherwise considered unstable by the investigator, based on medical history, physical examination, and routine laboratory tests.
* Patients who need to change or discontinue aspirin or clopidogrel, fail to take medication, or fail to come to the hospital on time due to their condition, and some information is missing.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic cardiovascular and cerebrovascular diseases in our hospital were included from January 2021 to December 2021, and from January 2021 to December 2021. All patients were male or female, aged ≥55 years.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding | MRI was used to assess bleeding at 180 ± 7 day and 360 ± 7 day. Cortical (lobar) hemorrhages were classified as microbleeds according to their size (<5 mm in diameter).
  MRI evaluated the degree and location of microbleeding

SECONDARY OUTCOMES:
Neurological symptom evaluation | Barthel index was measures at 6 and 12 months. With ten ordinally scaled items, functional status (dependency on nursing) of the patients is assessed (range from 0 is completely dependent on care to 100 is completely independent).
  Barthel index

IPD SHARING:
Plan to Share IPD: Undecided